CLINICAL TRIAL: NCT03409861
Title: Non-invasive, Non-Oscillometric Blood Pressure Band
Brief Title: 'Wristband Device for the Measurement of Intermittent Blood Pressure and Other Physiological Signals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: GuardLyff
Record Dates: First submitted 2018-01-03; First posted 2018-01-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A wristband device intended for use as a standalone device, designed for the measurement of intermittent blood pressure, as well as other physiological signals. The device is intended to be worn in day to day life by individuals suffering from hypertension or other conditions where monitoring of blood pressure is of importance.

DETAILED DESCRIPTION:
The device is intended to be worn on the wrist for intermittent measurements of vital signs such as HR, blood pressure, Skin temperature and activity.

The use does not require any special action from the user apart form wearing the band on either their left or right wrist. The device applies no inflatable mechanics or moving parts. The waistband is watertight and can be worn as any type of bracelet all the time of most of the time.

The study will focus on patients in intensive care or any other cardiology unit who are under continuous oversight of existing Invasive (A-line Gold Standard monitors

ELIGIBILITY:
Inclusion Criteria:

1. Signed written Institution approved Informed Consent Form (ICF)
2. Male and Females over the age of 18 years
3. Patients in intensive care or cardiology units who are under continuous oversight of existing Invasive (A-Line) Gold Standard monitors.
4. Only subjects who are fitted with an invasive Arterial Line (A LINE)
5. To the extent possible, individuals who have not been using medication 5 (five) hours prior to the test shall be classified as non-medicated subjects.

Exclusion Criteria:

1. Subject who are unable to provide consent
2. Where it would be impractical or inconvenient or otherwise unfeasible to place to place a wristband and generate a signal.
3. Subjects who are not fitted with, or not planned to be fitted with an A-Line during their stay in the hospital.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and females over the age of 18 years Patients who are already fitted with and invasive Arterial Line (A-Line)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Monitoring | 30-60 seconds of a clean signal from the A-line monitor
  Wearing of a non invasive wristband to measure Blood Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Shotan, Prof, Principal Investigator — Principal Investigator